CLINICAL TRIAL: NCT00660621
Title: A Phase II Study Of Gliadel, Concomitant Temozolomide And Radiation, Followed By Dose Dense Therapy With Temozolomide Plus Bevacizumab For Newly Diagnosed Malignant High Grade Glioma
Acronym: KARE004
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kentuckiana Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Renato V. LaRocca, MD, Kentuckiana Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KARE004; KARE004
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Glioma
Keywords: High Grade; Malignant; GBM
MeSH Terms: conditions — Glioma | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temozolomide and Bevacizumab — Between 14 and 28 days after surgery, all subjects will begin a standard course of post-operative limited field radiation therapy to the tumor site and a surrounding margin with concomitant temozolomide at a daily dose of 75 mg/m2 (7 days/week).
  No later than 45 days after date of completion of radiation therapy, all subjects will begin dose dense temozolomide at dose of 150 mg/m2 on Days 1-7 and 15-21 of a 28 day cycle with concomitant bevacizumab 10mg/kg administered intravenously every other week.

SUMMARY:
To determine the safety and efficacy of surgical resection with Gliadel® 3.85% wafer implantation, followed by concomitant limited field radiation therapy and temozolomide, followed by dose dense temozolomide and bevacizumab in subjects undergoing initial surgery for newly-diagnosed high grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, men and women, must be between ages 18 and 75 years.
* Subjects must have radiographic evidence on cranial magnetic resonance imaging (MRI) of a single, contrast-enhancing unilateral supratentorial cerebral tumor.
* Surgery is recommended within 4 weeks of the baseline MRI scan.
* Subjects must have a Karnofsky Performance Score of 60 or higher.
* Subjects must have signed an Institutional Review Board (IRB)-approved informed consent prior to any non-standard of care study procedure or no later than the start of dose dense temozolomide and bevacizumab..
* Subjects must have a pathological diagnosis of a high grade (IV) malignant glioma.
* Subjects, both men and women, must be willing to avoid pregnancy for up to 2 years after wafer implantation surgery and be counseled regarding the unknown, and potentially harmful, risks to the embryo or fetus from participation in this study.

Exclusion Criteria:

* Subjects who have had prior cytoreductive surgery for high-grade glioma. Subjects who have had a diagnostic stereotactic biopsy are eligible.
* Subjects with more than one focus of tumor or tumor crossing the midline as assessed by coronal cranial MRI scan.
* Concomitant significant life-threatening disease from which the subject could reasonably be expected to die within the first 12 months of the study.
* Known hypersensitivity reactions to temozolomide, nitrosoureas or any other components of the Gliadel® wafer.
* Prior CNS radiotherapy.
* Subjects who have received any prior chemotherapy for this malignant glioma prior to the baseline evaluation or subjects who are currently being treated with chemotherapeutic agents.
* Subjects with fewer than 100,000 platelets per mm3 or fewer than 3.500 leukocytes per mm3.
* Liver function tests greater than or equal to 2.5 times the upper limit of normal (transaminases (SGOT, SGPT), total bilirubin, alkaline phosphatase).
* Serum creatinine equal to or greater than 1.5 times the upper limit of normal, blood urea nitrogen (BUN) equal to or greater than 2.5 times the upper limit of normal.
* Pregnancy, or lactating females or females of childbearing potential not using adequate contraception.
* Participation in any other investigational protocol in the prior twelve months for any type of malignancy.
* Psychological, familial, sociological or geographical conditions which do not permit adequate medical follow-up and compliance with the study protocol.
* Inadequately controlled hypertension (blood pressure systolic > 150 mmHg or diastolic > 100 mmHg).
* Unstable angina or history of myocardial infarction within six months prior to enrollment.
* Evidence of bleeding, diathesis, or coagulopathy. Chronic full-dose anticoagulation with warfarin is not permitted though subjects may be on low molecular weight heparin or fondaparinux.
* Serious non-healing wound, ulcer, or bone fracture.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of concomitant limited field radiation therapy and temozolomide, followed by dose dense temozolomide and bevacizumab in subjects undergoing initial surgery for newly-diagnosed high grade glioma. | First 5 subjects after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Renato V. LaRocca, MD, Principal Investigator — Kentuckiana Cancer Instititue
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States